CLINICAL TRIAL: NCT04122651
Title: Randomised, Controlled Study Comparing Use of "Off the Shelf" Toric Lenses, With Set Cylindrical Corrections (2.00D or 4.00D) and Combined Limbal Relaxing Incisions and/or Off-axis Lens Rotation, With Fully Targeted Toric Lens Correction.
Brief Title: Toric Intraocular Lenses for Cataract Patients in the NHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 265865
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cataract; Astigmatism; Cornea
MeSH Terms: conditions — Cataract; Astigmatism; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Rayone Toric intraocular lens (for cataract surgery)
Who Masked: Participant
Masking Description: Patients will be randomised into one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Patients will be receiving a toric intraocular lens with either a 2.00 or 4.00 diopter (D) correction, depending on the degree of pre-operative astigmatism, and the astigmatic refractive error will be refined with the use of adjunctive limbal relaxing incisions LRIs and/or off axis rotation of the toric IOL (based on a standardized protocol) so the full amount of corneal astigmatism can be targeted for correction for each patient.
  Interventions: Procedure: 'Off the shelf' toric lens
- Control Arm (Active Comparator): The patient will receive a toric intraocular lens individually tailored to and ordered for each patients' precise degree of corneal astigmatism.
  Interventions: Procedure: Tailored Toric lens

INTERVENTIONS:
Procedure: 'Off the shelf' toric lens — 'Off the shelf' toric lens (either 2.00D or 4.00D) and combined limbal relaxing incisions and/or off-axis inttaocular lens rotation
  Arms: Experimental Arm
Procedure: Tailored Toric lens — Fully targeted toric intraocular lens correction for corneal astigmatism
  Arms: Control Arm

SUMMARY:
To assess visual performance, refractive outcome, and patient satisfaction with the use of "off the shelf" toric lenses, with a set cylindrical correction of 2.00 or 4.00 diopters, and combined limbal relaxing incisions and/or off-axis intraocular lens rotation, compared to fully targeted toric intraocular lens correction.

DETAILED DESCRIPTION:
The aim of this study is to evaluate a simplified, more cost-effective procedure for the use of toric intraocular lenses, with a focus on suitability for NHS cataract surgery. This study will involve the use of standard, "off-the-shelf" toric lenses rather than having them specifically tailored and ordered for each individual patient. Eligible participants (>1.25 D of corneal astigmatism) will be randomised, receiving a toric IOL with either a 2.00 or 4.00 diopter (D) correction, depending on the degree of pre-operative astigmatism, or a toric IOL individually tailored to and ordered for each patients' precise degree of corneal astigmatism. With the "off the shelf" toric IOL group the correction of the astigmatic refractive error will be refined with the use of adjunctive limbal relaxing incisions LRIs and/or off axis rotation of the toric IOL (based on a standardized protocol) so the full amount of corneal astigmatism can be targeted for correction for each patient. The clinical outcome will then be measured and compared between the 2 groups. Independent safety monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral or unilateral cataracts requiring surgical intervention
2. Age over 18 years
3. Able to understand informed consent and the objectives of the trial
4. Not pregnant, not breast feeding
5. No previous eye surgery
6. Corneal astigmatism greater than 1.5 diopters in one eye.

Exclusion Criteria:

1. age-related macula degeneration
2. glaucoma
3. previous retinal vascular disorders
4. previous retinal detachment or tear
5. any neuro-ophthalmological condition
6. any inherited retinal disorder or pathology
7. previous strabismus surgery or record of amblyopia
8. previous TIA, CVA or other vaso-occlusive disease
9. already enrolled in another study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-10-14 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Visual Acuities | 6 months
  Corrected and uncorrected Logmar Visual Acuities
Refractive Error | 6 months

SECONDARY OUTCOMES:
Intraoperative and post operative complications | 0 day-6 months
Patient Satisfaction | 6 months
  Patient satisfaction scores using validated questionnaires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naderi K, Jameel A, Chow I, Hull C, O'Brart D. Effects of axis-flip of the refractive cylinder on vision and patient-reported outcome measures after toric intraocular lens implantation. J Cataract Refract Surg. 2024 Dec 1;50(12):1230-1235. doi: 10.1097/j.jcrs.0000000000001530. PMID 39073343